CLINICAL TRIAL: NCT00224445
Title: Boosted Atazanavir and Truvada Given Once-Daily (BATON Study): A Phase 4 Study of Safety, Efficacy & Adherence in HIV Infected, Antiretroviral Naïve Subjects Treated With a Simple Once-Daily Regimen
Brief Title: Boosted Atazanavir and Truvada Given Once-Daily - BATON Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-164-0115
Record Dates: First submitted 2005-09-20; First posted 2005-09-23 (Estimated); Last update posted 2013-01-10 (Estimated); Status verified 2013-01

CONDITIONS: HIV Infections
Keywords: Treatment Naive; HIV-1
MeSH Terms: conditions — HIV Infections | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Atazanavir Sulfate; Ritonavir

ARMS (1):
- Truvada + Ritonavir-boosted Atazanavir (Experimental): All participants received Truvada plus ritonavir-boosted atazanavir
  Interventions: Drug: Truvada; Drug: Atazanavir; Drug: Ritonavir

INTERVENTIONS:
Drug: Truvada — Truvada (emtricitabine 200 mg/tenofovir disoproxil fumarate 300 mg tablet) administered orally once daily (QD)
Drug: Atazanavir — Atazanavir 300 mg (given as two 150-mg capsules) administered orally QD
Drug: Ritonavir — Ritonavir 100 mg capsule administered orally QD

SUMMARY:
To determine the safety and efficacy of a simple, once-daily antiretroviral (ARV) regimen consisting of a fixed-dose combination tablet containing Truvada combined with atazanavir boosted with ritonavir in treatment naive patients.

DETAILED DESCRIPTION:
To determine the safety and efficacy (viral load suppression and cluster of differentiation 4 [CD4] changes) of a simple, once-daily (QD) antiretroviral (ARV) regimen consisting of a fixed-dose combination tablet containing Truvada combined with the protease inhibitor atazanavir (ATV) boosted with ritonavir (ATV/r).

To evaluate fasting glucose, insulin, C peptide and lipid panel (total cholesterol, high and low density lipoprotein cholesterol (HDL, LDL), and serum triglycerides) in subjects receiving Truvada and boosted atazanavir.

To evaluate adherence to a QD ARV regimen of Truvada and boosted atazanavir.

To evaluate steady-state plasma pharmacokinetics (PK) of Truvada and atazanavir in study subjects receiving Truvada and boosted atazanavir.

ELIGIBILITY:
Inclusion Criteria:

* Adult (greater than or equal to 18 years) male or non-pregnant female HIV 1- infected subjects regardless of race or ethnicity.
* Antiretroviral treatment-naïve.
* Plasma HIV 1 RNA greater than 1000 copies/mL (Roche Amplicor HIV 1 Monitor Test Version 1.5 Ultrasensitive method, with a reflex to Standard for results greater than 75,000 and dilution for results greater than 750,000). There are no CD4 criteria for study inclusion.
* Adequate renal function defined as a calculated creatinine clearance (CLCr) greater than or equal to 50 mL/min according to the Cockcroft-Gault formula:
* Male: (140 - age in years) x (wt in kg) divided by 72 x (serum creatinine in mg/dL) = CLCr (mL/min.
* Female: (140 - age in years) x (wt in kg) divided by 72 x (serum creatinine in mg/dL) x 0.85 = CLCr (mL/min).
* Negative serum pregnancy test (females of childbearing potential only).
* Males and females (of childbearing potential, i.e. less than 2 years post-menopausal) must agree to avoid pregnancy by sexual abstinence, or utilization of a highly effective method of birth control throughout the study period and for 30 days following discontinuation of study drug.
* Life expectancy greater than or equal to 1 year.
* Subjects should be available for follow up for a period of at least 48 weeks.
* The ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures.

Exclusion Criteria:

* Prior antiretroviral treatment.
* Screening ALT greater than 5 x the upper limit of the normal range (ULN).
* Proven or suspected acute hepatitis in the 30 days prior to study entry. Subjects with chronic hepatitis are eligible provided that their liver transaminases (ALT) are less than 5 x ULN.
* A new AIDS defining condition diagnosed (with the exception of CD4 criteria) within 30 days of baseline.
* Previous therapy with agents with systemic myelosuppressive, pancreatoxic, hepatotoxic or cytotoxic potential within 3 months of study start or the expected need for such therapy at the time of enrollment.
* Presence of cardiomyopathy.
* Heart rate less than 40 bpm.
* Clinical symptoms potentially related to heart block (syncope, palpitations, unexplained dizziness)
* Known conduction disease.
* Third degree heart block.
* Clinically significant laboratory values that would preclude prescribing antiretroviral therapy, in the opinion of the investigator.
* Receiving ongoing therapy with any of the following (administration of any of the following medications must be discontinued at least 30 days prior to the Baseline visit and for the duration of the study period):

  * Nephrotoxic agents (aminoglycoside antibiotics, amphotericin B, cidofovir, cisplatin, foscarnet, IV pentamidine, other agents with significant nephrotoxic potential):
  * Adefovir dipivoxil
  * Probenecid
  * Systemic chemotherapeutic agents (i.e., cancer treatment medications)
  * Systemic corticosteroids
  * Interleukin 2 (IL 2)
  * Investigational agents (except upon approval by Gilead).
* Drugs that are contraindicated with atazanavir and/or ritonavir including:

  * midazolam
  * triazolam
  * ergot alkaloids
  * pimozide
  * proton-pump inhibitors
  * H2 blockers
  * lovastatin
  * simvastatin
  * diltiazem
  * amiodarone
  * bepridil
  * flecainide
  * propafenone
  * quinidine
  * St. John's Wort
  * rifampin
  * irinotecan
* Pregnant or lactating subjects.
* Evidence of a gastrointestinal malabsorption syndrome or chronic nausea or vomiting which may confer an inability to receive an orally administered medication.
* Current alcohol or substance abuse judged by the investigator to potentially interfere with subject adherence.
* Malignancy other than cutaneous Kaposi's sarcoma (KS) or basal cell carcinoma. Subjects with biopsy-confirmed cutaneous KS are eligible, but must not have received any systemic therapy for KS within 30 days of baseline and are not anticipated to require systemic therapy during the study.
* Active, serious infections (other than HIV 1 infection) requiring parenteral antimicrobial therapy within 15 days prior to screening.
* Prior history of significant renal or bone disease.
* Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the subject unsuitable for the study or unable to comply with the dosing requirements.
* Current imprisonment or involuntary incarceration in a medical facility for psychiatric or physical (e.g., infectious disease) illness.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2005-09; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Determine the safety/efficacy (viral load suppression and CD4 changes) of a once-daily (QD) antiretroviral (ARV) regimen consisting of a fixed-dose combination tablet containing Truvada. | Baseline to Week 48

SECONDARY OUTCOMES:
To evaluate fasting glucose, insulin, C peptide and lipid panel (total cholesterol, high and low density lipoprotein cholesterol (HDL, LDL), and serum triglycerides) in subjects receiving Truvada and boosted atazanavir. | Baseline to Week 48
To evaluate adherence to a QD ARV regimen of Truvada and boosted atazanavir. | Baseline to Week 48
To evaluate steady-state plasma PK of Truvada & atazanavir in study subjects receiving Truvada and boosted atazanavir. | Baseline to Week 48

CONTACTS AND LOCATIONS:
Overall Officials: John Flaherty, Study Director — Gilead Sciences
Locations (1):
- Gilead Sciences, Inc., Foster City, California, United States

REFERENCES:
- See also: Gilead Website — http://www.gilead.com
- See also: Truvada Website — http://www.truvada.com
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-US-164-0107_synopsis.pdf